CLINICAL TRIAL: NCT03175562
Title: A Human Repeat Insult Patch Test (HRIPT) in Healthy Subjects to Assess the Cutaneous Irritation and Sensitization Potential of a Cosmetic Facial Product
Brief Title: To Assess the Cutaneous Irritation and Sensitization Potential of a Cosmetic Facial Product Using a Human Repeat Insult Patch Test (HRIPT) in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 207585
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-06

CONDITIONS: Skin Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test product (Experimental): All the participants will have the test product applied to the appropriate test sites by trained study staff. The test site will be designated on above the waist between the left scapula and waistline and away from the spinal mid-line.
  Interventions: Other: Facial micellar cleanser
- Reference product (Other): All the participants will have the reference product applied to the appropriate test sites by trained study staff. The test site will be designated on above the waist between the left scapula and waistline and away from the spinal mid-line.
  Interventions: Other: Saline Solution: Sodium Chloride (NaCl; 0.9%)

INTERVENTIONS:
Other: Facial micellar cleanser — Participant will have each product applied topically via semi occlusive patch, on site by the technician. Each patch will remain in place for 48 (± 2) hours on weekdays and 72 (± 2) hours on weekends.
  Arms: Test product
Other: Saline Solution: Sodium Chloride (NaCl; 0.9%) — Participant will have each product applied topically via semi occlusive patch, on site by the technician. Each patch will remain in place for 48 (± 2) hours on weekdays and 72 (± 2) hours on weekends.
  Arms: Reference product

SUMMARY:
The objective of this clinical study is to assess the irritation and sensitisation potential of a cosmetic test product after repeated semi-occlusive patch applications to healthy human participants by following a conventional HRIPT methodology under supervision of a dermatologist.

DETAILED DESCRIPTION:
The first phase of the study is an Induction Phase; a known amount of each product (test and control) is applied, under a semi-occlusive patch. Patches will remain on the skin for 48 (±2) (weekdays) or 72 (±2) (including inclusive weekends) hours during this phase. Induction phase lasts for 3 weeks. After the Induction Phase participants will enter a Rest Phase of 2 weeks duration, during which no patches are applied. After the Rest Phase, participants will return to the clinical site for the Challenge Phase. In this phase a challenge patch containing the test and control products is applied to virgin skin for 48 (±2) hours then assessed 30 minutes (maximum 1 hour) following removal, 24 (± 2) and 48 (±2) hours later.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study procedures, restrictions and willingness to participate as evidenced by voluntary written informed consent and has received a signed and dated copy of the informed consent form
* Good general and mental health with, in the opinion of the investigator or medically qualified designee no clinically significant and relevant abnormalities in medical history or upon physical examination
* Healthy, intact skin at the proposed application site; dorsum (scapular region)
* Clinical assessment for eligibility (at Visit 1 and Visit 2 - if not combined) by a dermatologist to ensure participant is free of clinically relevant dermatological conditions
* Fitzpatrick phototype I to IV
* Agreement to comply with the procedures and requirements of the study and to attend the scheduled assessment visits

Exclusion Criteria:

* Women who are known to be pregnant or who are intending to become pregnant over the duration of the study
* Women who are breast-feeding
* Any history of significant dermatological diseases or conditions or medical conditions known to alter skin appearance or physiologic response (e.g. diabetes,) which could, in the opinion of the Investigator, preclude topical application of the investigational products and/or interfere with the evaluation of the test site reaction
* Presence of open sores, pimples, or cysts at the application site
* Active dermatosis (local or disseminated) that might interfere with the results of the study
* Considered immune compromised
* History of diseases aggravated or triggered by ultraviolet radiation
* Participants with dermatographism
* Currently using any medication which in the opinion of the investigator, may affect the evaluation of the study product, or place the participant at undue risk
* Use of the following topical or systemic medications: immunosuppressants, antihistamines, non-hormonal anti-inflammatory drugs, and corticosteroids up to 2 weeks before screening visit
* Oral or topical treatment with vitamin A acid and/or its derivatives up to 1 month before the screening visit
* Intention of being vaccinated during the study period or has been vaccinated within 3 weeks of the screening visit
* Currently receiving allergy injections, or received an allergy injection within 7 days prior to Visit 1, or expects to begin injections during study participation
* Previous history of atopy, allergic reactions, irritation or intense discomfort feelings to topical-use products, cosmetics or medication
* Study participants with a history of allergy to the study material/product, hypoallergenic tape, or to the cotton patches
* History of sensitisation in a previous patch study
* Participation in another clinical study (including cosmetic studies) or receipt of an investigational drug within 30 days of the screening visit
* Previous participation in this study
* Recent history (within the last 5 years) of alcohol or other substance abuse
* Intense sunlight exposure or sun tanning sessions up to 30 days before the Screening evaluation
* Intention of bathing (in the sea or a pool), sauna, water sports, or activities that lead to intense sweating
* Any participant who, in the judgment of the Investigator, should not participate in the study
* Any skin marks on the test site that might interfere with the evaluation of possible skin reactions (e.g. pigmentation disorders, vascular malformations, scars, tattoos, excessive hair, numerous freckles)
* Prisoner or involuntary incarcerated participant
* Participant from an indigenous tribe
* An employee of the sponsor or the study site or members of their immediate family

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2017-03-27 (Actual); Primary Completion 2017-05-19 (Actual); Study Completion 2017-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Valinhos, Brazil

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were enrolled at one center in Brazil.
Pre-assignment Details: A total of 294 participants were screened,out of which 240 participants were randomized and 54 participants were not randomized. Out of 54 participants, 22 participants did not meet study criteria, 5 participants were lost to follow-up, 26 participants withdrew their consent, 1 participant was not randomized for other reasons (not specified).
Groups:
- All Participants: Included all participants who were randomized to receive the study treatment. In this study, the test product and the negative control (saline solution) were randomly applied to 2 different cells in a single semi-occlusive patch that was applied on a subject's dorsum.
Period: Overall Study
Arm/Group | All Participants
Started | 240
Test Product (All participants received both the study treatments in a single semi-occlusive patch.) | 240
Negative Control (All participants received both the study treatments in a single semi-occlusive patch.) | 240
Completed | 224
Not Completed | 16
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 7
Not completed — Other (Not Specified) | 5

BASELINE CHARACTERISTICS:
Population: Safety population (N=240), the Safety population included all participants who received any application of the study products.
Groups:
- Overall Participants: All the participants who received any application of study products were included for baseline evaluation
Arm/Group | Overall Participants
Number analyzed (Participants) | 240
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.2 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196
  Male | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 234
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Induction Phase at Day 3
Description: A trained assessor assessed all patch sites. The following scores were used to express the response observed at the time of examination: 0=No evidence of irritation, 1=Minimal erythema; barely perceptible, 2=Definite erythema, readily visible; or minimal edema; or minimal papular response, 3=Erythema and papules, 4=Definite edema, 5=Erythema, edema, and papules, 6=Vesicular eruption, 7=Strong reaction spreading beyond test site. Other features indicative irritation (Superficial irritation) scores were: Grade A/Score 0=Slight glazed appearance, Grade B/Score 1=Marked glazing, Grade C/Score 2=Glazing with peeling and cracking, Grade F/Score 3=Glazing with fissures, Grade G/Score 3=Film of dried serous exudate covering all or portion of the patch, Grade H/Score 3=Small petechial erosions and/or scabs. Superficial irritation scores were only provided if there was a dermal response score >0. Full range was 0-10. Lower score indicates better tolerability.
Time Frame: At Day 3
Population: The Intent to treat (ITT, N=238) population included all participants who were randomized into the study and have skin irritation scores from at least one of the test sites available.
Measure: Mean (Standard Deviation); unit: Score on scale
Groups:
- Test Product: This arm included data from all the test sites were test product was applied.
- Reference Product: This arm included data from all the test sites were negative control was applied.
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 238 | 238
Score on scale | 0 (0) | 0 (0)

2. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Induction Phase at Day 5
Description: as for outcome 1
Time Frame: At Day 5
Population: The ITT (N=238) population included all participants who were randomized into the study and have skin irritation scores from at least one of the test sites available.
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 238 | 238
Score on scale | 0 (0) | 0 (0)

3. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Induction Phase at Day 8
Description: as for outcome 1
Time Frame: At Day 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 238 | 238
Score on scale | 0 (0) | 0 (0)

4. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Induction Phase at Day 10
Description: as for outcome 1
Time Frame: At Day 10
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 238 | 238
Score on scale | 0 (0) | 0 (0)

5. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Induction Phase at Day 12
Description: as for outcome 1
Time Frame: At Day 12
Population: as for outcome 2
Measure: Mean (Standard Error); unit: Score on scale
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 238 | 238
Score on scale | 0 (0) | 0 (0)

6. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Induction Phase at Day 15
Description: as for outcome 1
Time Frame: At Day 15
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 238 | 238
Score on scale | 0 (0) | 0 (0)

7. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Induction Phase at Day 17
Description: as for outcome 1
Time Frame: At Day 17
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 238 | 238
Score on scale | 0 (0) | 0 (0)

8. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Induction Phase at Day 19
Description: as for outcome 1
Time Frame: At Day 19
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Test Product | Reference Product
Number analyzed (Participants) | 238 | 238
Score on scale | 0 (0) | 0 (0)

9. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Challenge Phase at Week 6 After 30 Minutes (Maximum 1 Hour) Post Patch Removal
Description: as for outcome 1
Time Frame: At Week 6 after 30 minutes (maximum 1 hour) post patch removal
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on scale
Groups:
- Negative Control: This arm included data from all the test sites were negative control was applied.
Arm/Group | Test Product | Negative Control
Number analyzed (Participants) | 238 | 238
Score on scale | 0 (0) | 0 (0)

10. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Challenge Phase at Week 6 After 24 (±2) Hours Post Patch Removal
Description: as for outcome 1
Time Frame: At Week 6 after 24 (±2) hours post patch removal
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on scale
Groups:
- Reference Control: This arm included data from all the test sites were negative control was applied.
Arm/Group | Test Product | Reference Control
Number analyzed (Participants) | 238 | 238
Score on scale | 0 (0) | 0 (0)

11. Primary Outcome: Combined Skin Irritation (Dermal Response) and Superficial Irritation (Other Effects) Scores at Challenge Phase at 6 Week 48 (±2) Hours, Post Patch Removal
Description: as for outcome 1
Time Frame: At Week 6 after 48 (±2) hours post patch removal
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Test Product | Reference Control
Number analyzed (Participants) | 238 | 238
Score on scale | 0 (0) | 0 (0)

ADVERSE EVENTS:
Time Frame: Approximately 45 days
Groups:
- All Participants: Safety population (N=240), the Safety population included all participants who received any application of the study products.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/240
Serious Adverse Events (participants affected / at risk) | 0/240
Other Adverse Events (participants affected / at risk) | 6/240
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=240)
INFLUENZA (Infections and infestations) | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 1
TONSILLITIS BACTERIAL (Infections and infestations) | 1
VOMITING (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/62/NCT03175562/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-09): https://cdn.clinicaltrials.gov/large-docs/62/NCT03175562/SAP_001.pdf